CLINICAL TRIAL: NCT04126005
Title: A Combination Retrospective Medical History and Prospective Observational Study of Patients With Canavan Disease for Assessment of Natural History of Canavan Disease
Brief Title: Natural History Study of Patients With Canavan Disease (CANinform Study)
Status: Active, not recruiting | Type: Observational
Sponsor: Aspa Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: CVN-101; CANinform (Other: Aspa Therapeutics)
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2024-10

CONDITIONS: Canavan Disease
Keywords: Canavan Disease; AAV; AAV9; Gene therapy; Aspartoacylase; ASPA; ASPA gene; rAAV9; ACY2; Aminoacylase 2; Spongy degeneration; N-acetyl-L-aspartic acid (NAA); N-acetylaspartate; Rare disease; Inherited Metabolic Disorders; Leukodystrophy; Leukoencephalopathies; Autosomal Recessive Disorder; Neurodevelopmental diseases; CANinform Study
MeSH Terms: conditions — Canavan Disease; Rare Diseases; Leukoencephalopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Hematology, blood chemistry, urinalysis, genetic mutation confirmation, antibody testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Cohort 1 (Age < 18 Months): * Motor function assessments (remote or in-clinic) every 2 months
  * Clinic assessments every 6 months
- Cohort 2 (Age ≥ 18 Months - 3 Years): * Motor function assessments (remote or in-clinic) every 4 months
  * Clinic assessments every 6 months
- Cohort 3 (Age > 3 - 5 Years): * Motor function assessments (remote or in-clinic) every 6 months
  * Clinic assessments every 6 months
- Cohort 4 (Age > 5 Years): * Motor function assessments (remote or in-clinic) 12 months
  * Clinic assessments every 12 months
- Cohort 5 (Deceased): • The patient's medical history records will be reviewed. In addition, a parent interview will be performed.

SUMMARY:
This study uses medical records that allow retrospective data extraction of critical milestone and motor function data. In addition, prospective assessments collect data relevant to the natural history of Canavan disease in children.

DETAILED DESCRIPTION:
The CANinform natural history study is the first multinational effort to rigorously gather both retrospective and prospective data from this patient population. Data collection includes extraction of retrospective data from medical records of living and deceased patients, and collection of prospective, longitudinal data from living patients and their parent(s)/caregiver(s). Motor function assessments are performed remotely in the home via video or in the clinic by qualified study team members. Families will be invited to attend clinic visits and/or will be followed remotely by the clinical site for approximately 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Meet age criteria of a specific cohort.
2. Confirmed clinical and biochemical diagnosis of Canavan disease.
3. Available medical records since birth that permit documentation of disease characteristics and developmental milestones.
4. Parent and/or legal guardian is able to read, understand, and sign the informed consent.

Exclusion Criteria:

1. Patient does not meet the Inclusion Criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Living and deceased patients with Canavan disease
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
To characterize the natural history of Canavan disease | approximately 3 years
  To enhance the understanding of the natural history of Canavan disease through retrospective data collection from patient medical records and prospective data collection from living patients, including: phenotypic characteristics and variability, genotype characteristics and variability, and disease progression and natural history.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Massachusetts General Hospital, Boston, Massachusetts
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available for researchers using a defined process.

REFERENCES:
- See also: Aspa Therapeutics Company Website — http://aspatx.com
- See also: CANinform Study Website — http://treatcanavan.com